CLINICAL TRIAL: NCT02620553
Title: Primary Intervention With Mucosal Insulin for Prevention of Type 1 Diabetes in Infants at High Genetic Risk to Develop Diabetes POINT (Primary Oral Insulin Trial) A Dose Finding and Safety Study ( Pre-POINT )
Brief Title: Primary Intervention With Mucosal Insulin
Acronym: Pre-POINT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: University Hospital Dresden (Other); Diabetes Research Institute, Munich, Germany. (Unknown); University of Bristol (Other); Juvenile Diabetes Research Foundation (Other); German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 05-1043
Record Dates: First submitted 2015-06-08; First posted 2015-12-03 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; Diabetes; Autoimmune Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — Insulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Human Insulin (Experimental): Oral Insulin at 2.5 mg, 7.5 mg, 22.5 mg, or 67.5 mg per day
  Interventions: Drug: Human Insulin
- Placebo (Placebo Comparator): Oral Placebo
  Interventions: Other: Oral Placebo

INTERVENTIONS:
Drug: Human Insulin — There is a study drug dose increase once during the study. The dose increase will occur 6 months after entering into the study. A total of 6 children will be included at each dose (3 children will not have received insulin prior to entering the study and 3 children will have received a lower dose of insulin for 6 months). Further dose increases or more frequent dose increases in individual children will not be performed during Pre-POINT. Escalation will occur in both treatment and placebo group so that participants and study investigators will remain blinded to treatment throughout the study. First dose (2.5 mg oral insulin/day) Second dose (7.5 mg oral insulin/day) Third dose (22.5 mg oral insulin/day) Fourth dose (67.5 mg oral insulin/day)
  Other Names: Oral Insulin
  Arms: Human Insulin
Other: Oral Placebo — Oral Placebo is given orally daily
  Arms: Placebo

SUMMARY:
A dose with proven drug bioavailability to the immune system for use in a phase II/III primary T1DM (type 1 diabetes) vaccination trial (POINT study) in genetically at risk subjects.

Study Design Randomized, placebo-controlled, double-blind/double-masked, multi-center, dose escalation primary intervention pilot study.

Accrual Objective 25 (3:2 randomization to active and control arms)

DETAILED DESCRIPTION:
The objective of this study is to determine the feasibility, safety and bioavailability of oral insulin in children with high genetic risk for T1DM in a dose escalation primary intervention pilot study.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 2 years to 7 years who:

   * Have a multiplex first degree family history of T1DM (both parents, parent and sib, or two sibs);
   * Type 1 diabetes susceptible HLA DR4-DQB1*0302 or DR4-DQB1*0304 haplotype and

   None of the following HLA DR or DQB1 alleles:
   * DR 11
   * DR 12
   * DQB1*0602
   * DR7-DQB1*0303
   * DR14-DQB1*0503 or
   * Have a sibling with T1DM;
   * Identical by descent for the HLA DR3/DR4-DQ8 genotype with their diabetic sibling;
2. Islet autoantibody negative at time of recruitment.

Exclusion Criteria:

1. Children with any kind of congenital or acquired chronic disease that potentially interfere with the study objectives.
2. Prior or current participation in another intervention trial.
3. Chronic oral steroid use and/or other chronic oral immunosuppressant

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2007-09; Primary Completion 2013-06 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change in Blood Glucose Levels | Day 1
  Evaluation for hypoglycemia will be measured prior to administration of the insulin (baseline), then at 30, 60, and 120 minutes after administration of the insulin.
Daily Evaluation of Blood Glucose Levels | Days 2 through 7
  Blood glucose will be measured 60 minutes after the administration of the Insulin.
Evaluation of Blood Glucose Levels | Measured 60 minutes after oral insulin dosing, every day during each 4th week, as long as the subject is given oral insulin.
  After treatment day 7, Insulin will be administered and measured on a monthly basis.

SECONDARY OUTCOMES:
Change in Total IgE and IgE. | 2 weeks, 3 months, 6 months
  Allergy/intolerance to the study drug evaluated with total IgE and IgE antibodies to insulin at 2 weeks, 3 months, 6 months, then every 6 months thereafter, as well as monitored through self-reporting by families. Parents/guardians will be educated on and instructed to look out for possible allergic reactions to insulin.
T-cell responses related to potential immune response to Insulin | Day 1, 15 days, 3 and 6 months.
  T-cell responses e.g. antibody and cell mediated immune results will be evaluated the day of administration then at 15 days, 3 and 6 months, and every 6 months of treatment, and will be reported directly to the Data Coordinating Center.

CONTACTS AND LOCATIONS:
Overall Officials: Ezio Bonifacio, PhD, Principal Investigator — Medical Faculty Carl Gustav Carus, Dresden University of Technology; Georgeanna J Klingensmith, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Barbara Davis Center for Childhood Diabetes, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Bonifacio E, Ziegler AG, Klingensmith G, Schober E, Bingley PJ, Rottenkolber M, Theil A, Eugster A, Puff R, Peplow C, Buettner F, Lange K, Hasford J, Achenbach P; Pre-POINT Study Group. Effects of high-dose oral insulin on immune responses in children at high risk for type 1 diabetes: the Pre-POINT randomized clinical trial. JAMA. 2015 Apr 21;313(15):1541-9. doi: 10.1001/jama.2015.2928. PMID 25898052
- See also: Pre-POINT — http://www.diabetes-point.org/uk.html